CLINICAL TRIAL: NCT05082779
Title: A Phase I, Randomized, Double-Blind, Placebo-Contralled, Single Asending Dose / Multiple Ascending Dose Study of CS0159 to to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics, and Effect Food in Healthy Subject
Brief Title: Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CS0159
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascade Pharmaceuticals, Inc (Other)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0159-001
Record Dates: First submitted 2021-09-25; First posted 2021-10-19 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-10

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort A1: 0.2 mg (Experimental): Participants in fasted state will receive CS0159 0.2 mg or placebo once on Day 1.
  Interventions: Drug: CS0159
- Cohort A2: 0.6 mg (Experimental): Participants in fasted state will receive CS0159 0.6 mg or placebo once on Day 1.
  Interventions: Drug: CS0159
- Cohort A3: 1 mg (Experimental): Participants in fasted state will receive CS0159 1 mg or placebo once on Day 1 followed by a 7-day washout period then given in 1 mg tablet (in fed state) on Day 8.
  Interventions: Drug: CS0159
- Cohort A4: 2 mg (Experimental): Participants in fasted state will receive CS0159 2 mg or placebo once on Day 1.
  Interventions: Drug: CS0159
- Cohort A5: 4 mg (Experimental): Participants in fasted state will receive CS0159 4 mg or placebo once on Day 1.
  Interventions: Drug: CS0159
- Cohort A6: 8 mg (Experimental): Participants in fasted state will receive CS0159 8 mg or placebo once on Day 1.
  Interventions: Drug: CS0159
- Cohort B1: 0.4 mg (Experimental): Participants in fasted state will receive CS0159 0.4 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS0159
- Cohort B2: 1 mg (Experimental): Participants in fasted state will receive CS0159 1 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS0159
- Cohort B3: 2 mg (Experimental): Participants in fasted state will receive CS0159 2 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS0159
- Cohort B4: 4mg (Experimental): Participants in fasted state will receive CS0159 4 mg or placebo once daily for a consecutive 14 days.
  Interventions: Drug: CS0159

INTERVENTIONS:
Drug: CS0159 — Tablets administered orally
  Other Names: Placebo

SUMMARY:
The whole study includes 2 parts. Both the SAD study and MAD study are randomized, double-blinded, and placebo-controlled studies, conducted in healthy subjects, to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics profiles of CS0159. The SAD part also involves a pilot food effect (FE) study, designed to assess the food effect on single-dose PK profile in healthy subjects.

DETAILED DESCRIPTION:
A total of 48 healthy subjects will be allocated to 1 of 6 cohorts (cohort A1~A6) in the SAD study, each cohort including 8 subjects (6 subjects will receive investigational new drug (IND) product and 2 receive placebo). Each subject in fasted state will be randomly assigned to receive a single oral dose of CS0159 or placebo.To ensure the safety for all SAD cohorts (including A3 in both treatment periods).

The MAD study will enroll 32 healthy subjects, allocated to 1 of 4 cohorts (cohort B1~B4) and each cohort including 8 participants (6 subjects will receive IND products and 2 receive placebo). Subjects will be randomly assigned to orally receive the IND product or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant female volunteers
2. In good health, determined by having no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations

Exclusion Criteria:

1. Subjects with special dietary requirements and cannot follow a uniform diet.
2. Pregnant or nursing females or females who have pregnancy plans during the trial or within 3 months after the trial.
3. Any subject with SARS-CoV-2 infection, based on a positive polymerase chain reaction for SARS-CoV-2.
4. History or evidence of clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluations, procedures, or completion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Single-Dose Pharmacokinetic (PK) Parameter | Day 1 after dosing
  Area under the concentration-time curve (AUC) from time zero to infinity (AUC0-∞)
Single-Dose Pharmacokinetic (PK) Parameter: (AUC0-last) | Day 1 after dosing
  AUC from time zero to the time of the last measured concentration
Single-Dose Pharmacokinetic (PK) Parameter: (Cmax) | Day 1 after dosing
  Maximum observed plasma concentration
Single-Dose Pharmacokinetic (PK) Parameter: (Tmax) | Day 1 after dosing
  Time of the maximum observed plasma concentration
Multiple-Dose PK Parameter | Day 1 after dosing; day 14
  Maximum concentration during a dosing interval Ct_max
Multiple-Dose PK Parameter: (Ct_min, Day 14) | Day 1 after dosing; day 14
  Minimum concentration during a dosing interval
Multiple-Dose PK Parameter: (AUCtau) | Day 1 after dosing; day 14
  AUC over one dosing interval
To characterize the safety and tolerability of single dose of CS0159 | up to Day 31
  Incidence and severity of adverse events
To characterize the safety and tolerability of multiple doses of CS0159 | up to Day 44
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacodynamic (PD) Parameter: FGF19 | Day -1; day 1
  fibroblast growth factor 19
Pharmacodynamic (PD) Parameter: C4 | Day -1; day 1
  serum concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Doisy, MD, Principal Investigator — Labcorp Clinical Research Unit, Inc.
Locations (1):
- Labcorp Clinical Research Unit, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No